CLINICAL TRIAL: NCT03280264
Title: An Intra-Subject Dose-Adjustment Study of KHK7580 for the Treatment of Hypercalcemia in Patients With Parathyroid Carcinoma or Primary Hyperparathyroidism Who Are Unable to Undergo Parathyroidectomy or Relapse After Parathyroidectomy
Brief Title: Phase 3 Study of KHK7580 for the Treatment of Hypercalcemia in Patients With Parathyroid Carcinoma or Primary Hyperparathyroidism
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7580-101
Record Dates: First submitted 2017-09-07; First posted 2017-09-12 (Actual); Results first posted 2021-05-27 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Parathyroid Carcinoma; Primary Hyperparathyroidism
MeSH Terms: conditions — Parathyroid Neoplasms; Hyperparathyroidism, Primary | interventions — evocalcet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KHK7580 (Experimental): oral administration
  Interventions: Drug: KHK7580

INTERVENTIONS:
Drug: KHK7580 — oral administration
  Other Names: evocalcet

SUMMARY:
To evaluate the efficacy of KHK7580 orally administered up to 24 weeks for hypercalcemia in patient with parathyroid carcinoma or primary hyperparathyroidism who are unable to undergo parathyroidectomy or relapse after parathyroidectomy.

ELIGIBILITY:
Inclusion Criteria:

* Personally submitted written voluntary informed consent to participate in the study
* Patients with a diagnosis of parathyroid carcinoma or primary hyperparathyroidism who are unable to undergo parathyroidectomy or relapse after parathyroidectomy.
* Corrected serum calcium level is > 11.3 mg/dL at screening.

Exclusion Criteria:

* Patients receiving cinacalcet hydrochloride within 2 weeks before screening
* Patients diagnosed with hypercalcemia associated with malignant tumors other than parathyroid carcinoma.
* Severe heart disease
* Severe hepatic dysfunction
* Uncontrolled hypertension and/or diabetes
* Treatment with an investigational product (drug or medical device) in a clinical study or any study equivalent to clinical study within 12 weeks before screening

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2019-04-09 (Actual); Study Completion 2019-04-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Osaka City University Hospital, Ōsaka, Japan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- KHK7580 (2-24 mg): KHK7580 was orally administered daily for up to week 52.
Period: Overall Study
Arm/Group | KHK7580 (2-24 mg)
Started | 18
Completed | 15
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | KHK7580 (2-24 mg)
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 18
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 18
serum corrected Ca conc. [Mean (Standard Deviation); unit: mg/dL] | 11.73 (0.84)
serum intact Parathyroid Hormone conc. [Mean (Standard Deviation); unit: pg/mL] | 507.7 (1409.8)
parathyroid carcinoma [Count of Participants; unit: Participants] | 3
Unable to undergo parathyroidectomy [Number; unit: participants] | 13
Relapse after parathyroidectomy [Number; unit: participants] | 2
previous cinacalcet use [Number; unit: participants] | 13
Pharmacotherapy for primary diseases [Number; unit: participants] | 3
parathyroidectomy [Number; unit: participants] | 6
Parathyroid intervention therapy [Number; unit: participants] | 0

OUTCOME MEASURES:

1. Primary Outcome: The Number and Percentage of Patients Who Achived a Serum Corrected Ca Concentration of Under 10.3 mg/dL for at Least 2weeks During Titration Phase.
Time Frame: Up to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | KHK7580 (2-24 mg)
Number analyzed (Participants) | 18
Participants | 14

2. Secondary Outcome: The Number and Percentage of Patients in Whom the Decrease in Serum Corrected Ca Concentration From the Baseline Was ≥ 1.0 mg/dL for ≥ 2 Weeks During the Titration Phase.
Time Frame: up to 24 weeks
Measure: Count of Participants; unit: Participants
Groups:
- KHK7580 (2-24 mg): KHK7580 was orally administered daily.
Arm/Group | KHK7580 (2-24 mg)
Number analyzed (Participants) | 18
Participants | 12

3. Secondary Outcome: Serum Corrected Ca Level
Time Frame: up to 52 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | KHK7580 (2-24 mg)
Number analyzed (Participants) | 18
mg/dL | 9.89 (0.60)

4. Secondary Outcome: Serum Intact Parathyroid Hormone Level
Time Frame: up to 52 weeks
Measure: Mean (Standard Deviation); unit: pg/dL
Arm/Group | KHK7580 (2-24 mg)
Number analyzed (Participants) | 18
pg/dL | 152.6 (97.3)

5. Secondary Outcome: Serum Whole Parathyroid Hormone Level
Time Frame: up to 52 weeks
Measure: Mean (Standard Deviation); unit: pg/dL
Arm/Group | KHK7580 (2-24 mg)
Number analyzed (Participants) | 18
pg/dL | 108.9 (73.0)

ADVERSE EVENTS:
Time Frame: up to 52week
Arm/Group | KHK7580 (2-24 mg)
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 3/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | KHK7580 (2-24 mg) (N=18)
enterocolitis (Gastrointestinal disorders) | 1
urinary tract infection (Renal and urinary disorders) | 1
uterine cancer (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | KHK7580 (2-24 mg) (N=18)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cataract (Eye disorders) | 1
Cataract cortical (Eye disorders) | 1
Ocular hyperaemia (Eye disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain lower (Gastrointestinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Faeces soft (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 2
Hangover (General disorders) | 1
Nasopharyngitis (Infections and infestations) | 7
Cystitis (Infections and infestations) | 2
Influenza (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Hordeolum (Infections and infestations) | 1
Otitis externa (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Heat stroke (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1
Radiation sickness syndrome (Injury, poisoning and procedural complications) | 1
Blood creatinine increased (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-30): https://cdn.clinicaltrials.gov/large-docs/64/NCT03280264/Prot_SAP_000.pdf